CLINICAL TRIAL: NCT04306952
Title: Mind-Body Approach to Improve Health-Related Quality of Life for People With Narcolepsy
Brief Title: Awareness and Self-Compassion Enhancing Narcolepsy Treatment
Acronym: ASCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Mundt, PhD, Assistant Professor, Department of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00209890; R34AT009551 (NIH)
Record Dates: First submitted 2020-02-28; First posted 2020-03-13 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Narcolepsy; Narcolepsy Without Cataplexy; Narcolepsy With Cataplexy
Keywords: Narcolepsy; psychosocial; mindfulness; health-related quality of life; hypersomnia
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive one of there different MBI treatments: 1) Brief MBI, 4 weeks, 2) Standard MBI, 8 weeks, 3) Extended MBI, 12 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief MBI (Experimental): The brief MBI consists of four weekly group sessions that are two hours each and one all day mediation retreat.
  Interventions: Behavioral: Brief MBI
- Standard MBI (Experimental): The standard MBI consists of eight weekly group sessions that are approximately two hours each and one all day meditation retreat.
  Interventions: Behavioral: Standard MBI
- Extended MBI (Experimental): The extended MBI consists of four weekly group sessions followed by four group sessions every other week over the course of 12 weeks, with optional "office hours"in between the bi-weekly group sessions and one all day meditation retreat.
  Interventions: Behavioral: Extended MBI

INTERVENTIONS:
Behavioral: Brief MBI — The brief MBI consists of four weekly group sessions that are two hours each and one all day mediation retreat. The rationale for testing the short MBI is to evaluate a low-dose (8 hours of contact) MBI that optimizes cost-effectiveness and minimizes patient burden.
  Arms: Brief MBI
Behavioral: Standard MBI — The standard MBI consists of eight weekly group sessions that are approximately two hours each and one all day meditation retreat. The length of this package is based on the standard length of MBSR as an 8-week program. The rationale for testing the standard MBI is to provide a comparison to a dose (16 hours of contact) that is most similar to the length of MBSR and has the fewest modifications, making it easier to train MBI providers.
  Arms: Standard MBI
Behavioral: Extended MBI — The extended MBI consists of four weekly group sessions followed by four group sessions every other week over the course of 12 weeks. Each group session will be two hours. The group sessions will be identical to the standard package except for the timing (every other week) of the last four sessions. In addition to the group sessions, the MBI provider will offer "office hours" in between the bi-weekly group sessions, where participants will be able to schedule individual sessions with the MBI provider to discuss questions and troubleshoot their mindfulness practice. In addition, participants will receive an all-day meditation retreat, similar to the other conditions. The rationale for testing the extended MBI is to optimize acceptability and uptake based on the investigator's preliminary data by allowing for a slower, extended pace of learning mindfulness practices with an opportunity to have individual discussions with the instructor (16 hours of contact + individual office hours).
  Arms: Extended MBI

SUMMARY:
The overall goal of this research is to test the effectiveness of a mindfulness-based intervention (MBI) for improving health-related quality of life as a complementary practice to standard care for narcolepsy. This study is a feasibility trial in which 60 adults with narcolepsy will be randomized to receive either a 4-week (brief), 8-week (standard), or 12-week (extended) MBI. Each MBI will be delivered in small groups using a live videoconferencing platform and teaches mindfulness practices to help cope with narcolepsy symptoms. By developing a scalable mind-body intervention, this project can addresses a major research gap on improving psychosocial functioning in people with narcolepsy.

DETAILED DESCRIPTION:
Narcolepsy is a serious and debilitating condition involving persistent and excessive sleepiness that affects 1 in 2000 Americans and 3 million people worldwide. Although wake-promoting pharmacotherapy can reduce sleepiness there is no cure and people with narcolepsy experience significantly poor health-related quality of life, particularly in the domains of mental and social health. Therefore, the overarching goal of this research is to test the effectiveness of a mindfulness-based intervention (MBI) for improving health-related quality of life as a complementary practice to standard care for narcolepsy. The purpose of this study is to conduct a feasibility trial to determine the optimal parameters for adapting and delivering MBI to people with narcolepsy. The specific aims are to: 1) Determine the feasibility and acceptability of MBI delivered using videoconferencing for the purpose of improving psychosocial functioning in people with narcolepsy and 2) Determine the feasibility of recruitment and assessment methods for delivering MBI using videoconferencing. The feasibility trial includes 60 adults with narcolepsy who will be randomized to receive either a 4-week (brief), 8-week (standard), or 12-week (extended) MBI. Each MBI will be similar in content, which includes mindfulness practices and group discussions with adaptations for working with narcolepsy symptoms. All MBIs will be delivered in small groups using a live videoconferencing platform to enhance accessibility. If the findings of this project support the feasibility of further testing, the next project would be aimed at enhancing rigor and reproducibility (e.g., designing appropriate control, refining outcome measures and eligibility criteria) in preparation for a large-scale pragmatic trial. The overall significance of this research is to develop a scalable mind-body intervention that addresses a major research gap on improving psychosocial functioning in people with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18 and older (except when the age of majority for a state differs from 18, including Delaware [19 years or older], Mississippi [21 years or older], and Nebraska [19 years or older])
2. ICSD-3 criteria (8) for Narcolepsy (Type I or II)
3. Endorse current psychological distress based on a t-score ≥ 60 on the PROMIS depression or anxiety scales
4. Established standard care for narcolepsy. Patients who have not been previously diagnosed will be required to complete a clinical work-up through a sleep clinic (i.e., nocturnal PSG followed by a next-day MSLT) before participating. Standard care is managed outside of the study.

Exclusion Criteria:

1. Hypersomnia not of central origin (i.e., hypersomnia attributed to psychiatric disorder, medical disorder, other sleep disorder such as circadian rhythm sleep disorder, or insufficient sleep).
2. Current suicidal ideation or intent.
3. Uncontrolled medical conditions or physical limitations that require immediate medical treatment that would prevent ability to engage in the treatment protocol.
4. Inability to engage in the treatment protocol due to a psychiatric (e.g., psychotic disorder) or cognitive issue.
5. Untreated moderate-to-severe sleep-related breathing disorder, defined as an apnea hypopnea index (AHI) ≥ 15. Those receiving treatment for a sleep-related breathing disorder and can demonstrate adequate management (e.g., residual AHI < 5) will be allowed to participate.
6. Previous participation in a formal MBI program, such as MBSR.
7. Unstable dose of medications at the time of screening (e.g., stimulants).
8. Unable to attend intervention sessions due to accessibility (i.e., reliable internet connection) or availability (i.e., not available due to scheduling conflicts).
9. Currently living outside of the United States.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mundt, PhD, Principal Investigator — Northwestern University
Locations (1):
- Center for Circadian and Sleep Medicine, Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mundt JM, Zee PC, Schuiling MD, Hakenjos AJ, Victorson DE, Fox RS, Dawson SC, Rogers AE, Ong JC. Development of a mindfulness-based intervention for narcolepsy: a feasibility study. Sleep. 2024 Oct 11;47(10):zsae137. doi: 10.1093/sleep/zsae137. PMID 38895897

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Started | 20 | 20 | 20
Completed | 20 | 16 | 19
Not Completed | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief MBI | Standard MBI | Extended MBI | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 18 | 57
  >=65 years | 0 | 1 | 2 | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 16 | 17 | 20 | 53
  Male | 3 | 2 | 0 | 5
  Non-binary | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 18 | 18 | 18 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 18 | 20 | 17 | 55
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Patient-Reported Outcomes Measurement Information System Depression [Mean (Standard Deviation); unit: T-Score] — Measures depressive symptoms. Higher score indicates more depressive symptoms (worse outcome). Population mean (T-score) of 50 with a standard deviation of 10.
  T-Score | 59.53 (4.76) | 56.11 (4.81) | 60.06 (6.25) | 58.57 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Attended ≥ 80% of Sessions
Description: Number of participants who attended greater than or equal to 80% of sessions
Time Frame: 4 weeks (Brief MBI), 8 weeks (Standard MBI), or 12 weeks (Extended MBI)
Measure: Count of Participants; unit: Participants
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
Participants | 15 | 13 | 15

2. Primary Outcome: Number of Participants Who Practiced Meditation ≥ 4 Days Per Week
Description: Number of participants who practiced meditation greater than or equal to 4 days per week
Time Frame: 4 weeks (Brief MBI), 8 weeks (Standard MBI), or 12 weeks (Extended MBI)
Measure: Count of Participants; unit: Participants
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
Participants | 16 | 8 | 13

3. Primary Outcome: Number of Participants Who Completed Assessments
Description: Number of participants who completed entire baseline and post-treatment assessment (questionnaires, actigraphy, and neurocognitive testing)
Time Frame: Baseline and 4 weeks (Brief MBI), 8 weeks (Standard MBI), or 12 weeks (Extended MBI)
Measure: Count of Participants; unit: Participants
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
Participants | 18 | 13 | 16

4. Secondary Outcome: Self-Compassion Scale (SCS)
Description: The SCS assesses the acquisition of self-compassion. It is a 26-item self report measure with three main components of self-compassion: self-kindness vs. self-judgement, common humanity vs. isolation, and mindfulness vs. over-identification. The total score ranges from 1-5, with higher scores reflecting more self-compassion.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
score on a scale
  Baseline | 2.66 (.80) | 2.91 (.82) | 2.52 (.50)
  Post-treatment: number analyzed (Participants) | 19 | 18 | 17
  Post-treatment | 3.12 (.86) | 3.58 (.58) | 3.61 (.61)

5. Secondary Outcome: Five Facet Mindfulness Questionnaire (FFMQ)
Description: The FFMQ assesses the acquisition of mindfulness skills. It is a 39-item self-report measure that consists of five factors representing elements of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Total scores range from 39-195, with higher scores reflecting more mindfulness.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
score on a scale
  Baseline | 115.90 (24.80) | 122.50 (22.13) | 107.00 (13.43)
  Post-treatment: number analyzed (Participants) | 19 | 18 | 17
  Post-treatment | 132.42 (21.91) | 144.00 (16.11) | 136.53 (19.42)

6. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Psychosocial Illness Impact Positive
Description: Measures the direct positive psychosocial effect related to illness with higher scores reflecting better outcomes. Population mean (T-score) of 50 with a standard deviation of 10.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
T-score
  Baseline | 39.35 (8.00) | 42.07 (6.84) | 38.74 (7.23)
  Post-treatment: number analyzed (Participants) | 19 | 18 | 17
  Post-treatment | 42.83 (8.92) | 46.94 (8.26) | 43.85 (9.02)

7. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Psychosocial Illness Impact Negative Scale
Description: Measures the direct negative psychosocial effect related to illness with higher scores reflecting worse outcomes. Population mean (T-score) of 50 with a standard deviation of 10.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
T-score
  Baseline | 60.94 (6.53) | 59.35 (5.28) | 62.59 (8.26)
  Post-treatment: number analyzed (Participants) | 19 | 18 | 17
  Post-treatment | 58.70 (10.09) | 56.52 (6.24) | 57.28 (6.75)

8. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale
Description: Measures overall physical and mental health with higher scores reflecting better outcomes. Population mean (T-score) of 50 with a standard deviation of 10.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
T-score
  Global Mental Health (Baseline) | 38.01 (7.89) | 40.43 (6.07) | 36.03 (7.82)
  Global Mental Health (Post-treatment): number analyzed (Participants) | 19 | 18 | 17
  Global Mental Health (Post-treatment) | 41.17 (10.09) | 44.77 (7.35) | 42.73 (8.09)
  Global Physical Health (Baseline) | 46.32 (7.46) | 43.85 (6.15) | 43.71 (6.44)
  Global Physical Health (Post-treatment): number analyzed (Participants) | 19 | 18 | 17
  Global Physical Health (Post-treatment) | 47.41 (8.16) | 46.32 (6.82) | 45.12 (8.32)

9. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale
Description: Measures anxiety symptoms using Computer Adaptive Testing (CAT) with higher scores reflecting more anxiety symptoms (worse outcome). Population mean (T-score) of 50 with a standard deviation of 10.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
T-score
  Baseline | 62.54 (7.04) | 61.24 (4.85) | 61.69 (6.67)
  Post-treatment: number analyzed (Participants) | 19 | 18 | 17
  Post-treatment | 62.46 (9.79) | 56.62 (6.25) | 58.04 (7.48)

10. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Depression Scale
Description: Measures depressive symptoms using Computer Adaptive Testing (CAT) with higher scores reflecting more depressive symptoms (worse outcome). Population mean (T-score) of 50 with a standard deviation of 10.
Time Frame: Baseline to post-treatment (Brief MBI 4 weeks, Standard MBI 8 weeks, Extended MBI 12 weeks)
Population: Post-treatment scores not available for participants who did not complete the assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Brief MBI | Standard MBI | Extended MBI
Number analyzed (Participants) | 20 | 20 | 20
T-score
  Baseline | 59.53 (4.76) | 56.11 (4.81) | 60.06 (6.25)
  Post-treatment: number analyzed (Participants) | 19 | 18 | 17
  Post-treatment | 57.70 (9.08) | 53.89 (6.30) | 52.73 (6.08)

ADVERSE EVENTS:
Time Frame: 12 weeks (all groups)
Arm/Group | Brief MBI | Standard MBI | Extended MBI
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 5/20 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief MBI (N=20) | Standard MBI (N=20) | Extended MBI (N=20)
Stent placement (Cardiac disorders) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief MBI (N=20) | Standard MBI (N=20) | Extended MBI (N=20)
Actigraphy-related skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Exacerbation of pre-existing depression (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Car accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Increased sleepiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Melanoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT04306952/Prot_SAP_000.pdf